CLINICAL TRIAL: NCT00152633
Title: Effect of Losartan on Retinal Endothelial Function in Patients With Essential Hypertension
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No patient could be recruited.
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Retina-Losartan
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension
Keywords: endothelium, hypertension, retina, AT1
MeSH Terms: conditions — Hypertension | interventions — Losartan; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan (Active Comparator): Treatment with Losartan.
  Interventions: Drug: Losartan
- Betablocker (Active Comparator): Treatment with Metoprolol.
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Losartan
  Arms: Losartan
Drug: Metoprolol
  Arms: Betablocker
Drug: Losartan — Treatment with Losartan
  Arms: Losartan

SUMMARY:
Essential hypertension is commonly associated with impaired endothelial function. The retinal vasculature is morphologically and functionally related to the cerebral vessels because of the common origin from the internal carotid artery. A recent study in hypertensive patients demonstrated that endothelial function of the retinal vasculature is impaired in hypertensive patients and that it can be restored by treatment with an AT1-receptor antagonist. It is not clear whether this effect is due to blood pressure lowering or whether this is a blood pressure independent effect. The present randomized, double blind study with a cross over design addresses this issue by comparing the effects of losartan and metoprolol on retinal endothelial function in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65 years with essential hypertension

Exclusion Criteria:

* Secondary forms of hypertension
* Advanced damage of vital organs (grade III and IV retinopathy)
* History of serious hypersensitivity reaction to AT1-receptor blockers
* Actual or anamnestic alcohol- or drug abuse.
* Smokers or ex-smokers < 1 year.
* Patients with Diabetes mellitus (oral medication or insulin).
* Patients with arterial fibrillation or AV-Block (II° or more).
* Patients with anamnestic myocardial infarction.
* Patients with instable angina pectoris including EcG-aberrations or cardiac insufficiency NYHA III or IV.
* History of malignancy (unless a documented disease-free period exceeding 10 years is present) with teh exception of basal cell carcinoma of the skin
* History of allograft transplantation
* Therapy with not approved concomitant medication, or participation in a clinical study within 4 weeks preceding treatment start.
* Disease which interfere with the pharmacodynamics and pharmacokinetics of the study drug.
* Liver-or kidney disease with SGOT, GPT, g-GT, AP, bilirubin and creatinin or above 200% of standard.
* Patients, who are not sufficiently compliant, or patients, who are not capable or willing to appear for controlling vistas.
* Presumed risk of transmission of HIV or hepatitis via blood from the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change in retinal endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — CRC, Med. Klinik 4, University of Erlangen-Nürnberg
Locations (1):
- CRC, Med. Klinik 4, University of Erlangen-Nürnberg, Erlangen, Germany